CLINICAL TRIAL: NCT07160595
Title: Benefit on Chronic Pain of Early Screening and Management of Patients With Persistent Postoperative Pain at 3 Months
Acronym: DROPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 731_DROPS; ID RCB (Other: 2025-A01249-40)
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Chronic Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This study is a cluster crossover randomized trial. All participating centers (n=16) will take part in two sequential study periods:
  * Control Period: "Without early treatment at 3 months" During this period, patients with persistent postoperative pain-identified via SMS-will receive treatment at 6 months. This reflects the current standard of care for patients with postoperative pain.
  * Intervention Period: "With early treatment at 3 months" During this period, patients with persistent postoperative pain-identified via SMS-will receive early treatment starting at 3 months.
  Each center will be randomized into one of two sequences: "control period followed by intervention period" or "intervention period followed by control period."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control period 'without early intervention at 3 months' (No Intervention): During this period, patients with persistent post-operative pain, identified through SMS screening, will be treated at 6 months (this reflects the current standard experience for patients with postoperative pain).
- Intervention period 'with early intervention at 3 months' (Experimental): During this period, patients with persistent post-operative pain, identified through SMS screening, will receive early treatment starting at 3 months.
  Interventions: Other: Early management of postoperative pain at 3 months detected using sms

INTERVENTIONS:
Other: Early management of postoperative pain at 3 months detected using sms — During this period, patients with persistent post-operative pain, identified through SMS screening, will receive early treatment starting at 3 months.
  Arms: Intervention period 'with early intervention at 3 months'

SUMMARY:
Chronic postoperative pain has an overall incidence of approximately 30%, with 5% to 10% of cases classified as severe (numerical rating scale > 6/10). However, its management remains suboptimal, primarily due to underdiagnosis and delayed referral of patients to specialized chronic pain centers.

Improving the screening of patients with chronic postoperative pain is therefore crucial. Our research has shown that early detection of postoperative neuropathic pain is possible using just two text messages (SMS), as early as three months after surgery. Early screening, combined with prompt management, can prevent pain from becoming chronic and mitigate its harmful effects.

Study design

This study is a cluster crossover randomized trial. All participating centers (n=16) will take part in two sequential study periods:

* Control Period: "Without early treatment at 3 months" During this period, patients with persistent postoperative pain-identified via SMS-will receive treatment at 6 months. This reflects the current standard of care for patients with postoperative pain.
* Intervention Period: "With early treatment at 3 months" During this period, patients with persistent postoperative pain-identified via SMS-will receive early treatment starting at 3 months.

Study Population

The study will include patients undergoing the following minor surgical procedures:

* Inguinal hernia repair
* Breast reduction
* Mastectomy with lymph node dissection
* Knee arthroscopy
* Knee ligament reconstruction

Study Schedule Recruitment Period: 24 months Patient Follow-up: 6 months Total Estimated Study Duration: 30 months

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone one of the following procedures:

  * Inguinal hernia repair, regardless of the surgical technique used
  * Breast reduction
  * Mastectomy with or without reconstruction but with lymph node dissection
  * Knee arthroscopy or knee ligamentoplasty

    * Patients with a smartphone
    * French-speaking patients
    * Patients affiliated with a social security
    * Patients who have given their free and informed verbal consent

Exclusion Criteria:

* Patients with pain sensitivity defined by the presence of chronic pain, use of level 3 morphine analgesics, use of anxiolytics, gabapentinoids and/or antidepressants
* Patients subject to legal protection measures
* Patients deprived of their liberty
* Pregnant, labouring or breastfeeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2052 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with chronic post-operative pain at 6 months. | 6 months post-operative

SECONDARY OUTCOMES:
Types of chronic post-operative pain at 3 and 6 months: frequency of neuropathic pain and pain due to excessive nociception | 3 and 6 months post-operative
Proportion of patients responding to SMS during the various assessments | 3 and 6 months post-operative
Sensitivity and specificity of SMS for diagnosing pain with neuropathic characteristics post-operatively at 3 and 6 months | 3 and 6 month post-operative
Proportion of patients with pain at 3 and 6 months according to the type of surgery | 3 and 6 months post-operative

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - Hôpital Prive Claude Galien, Boussy-Saint-Antoine
  - Hospices Civils de Lyon, Lyon
  - Clinique Jules Verne, Nantes
  - Hôpital Privé du confluent Santé Atlantique, Nantes
  - AP-HP : Hôpital de la Pitié Salpêtrière, Paris
  - AP-HP : Hôpital Saint-Louis, Paris
  - Clinique Drouot Remusat, Paris
  - Clinique Geoffroy Saint Hilaire, Paris
  - Hôpital de la Croix Saint-Simon, Paris
  - Hôpital Paris Saint-Joseph, Paris
  - Institut Curie : Hôpital de Paris, Paris
  - Institut Mutualiste Montsouris, Paris
  - Institut Curie : Hôpital de Saint Cloud, Saint-Cloud
  - CHU de Saint-Etienne, Saint-Etienne
  - Hôpital Foch, Suresnes
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No